CLINICAL TRIAL: NCT04381325
Title: Phase I Clinical Trial to Evaluate the Safety and Tolerability and Pharmacokinetics of MSB0254 Injection in Patients With Advanced Solid Tumors
Brief Title: A Study of MSB0254 Injection in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Suzhou Transcenta Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSB0254-CSP-001
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSB0254 Injection (Experimental): This experiment will start from 4mg/kg with a dose increase of 3+3, and is planned to be carried out in 5 dose groups, namely 4mg/kg, 8mg/kg (100% increase), 12mg/kg (50% increase), 16mg/kg (33% increase) and 20mg/kg (25% increase).MSB0254 injection was administered intravenously on day 1 and day 15 every 28 days.To collect pharmacokinetic blood samples after repeated administration, MSB0254 injection was not administered on day 1 of the third cycle (C3D1).The observation period of DLT was 28 days after the first administration. An intravenous infusion with concentration 20 mg/kg every 3 weeks (Q3W).
  Interventions: Drug: MSB0254 Injection

INTERVENTIONS:
Drug: MSB0254 Injection — An intravenous infusion with concentration from 4 mg/kg to 16 mg/kg every 2 weeks (Q2W).
  An intravenous infusion with concentration 20 mg/kg every 3 weeks (Q3W).

SUMMARY:
This study was an open, multi-dose dose escalation phase I clinical study to evaluate the safety, tolerability and PK characteristics of MSB0254 in patients with locally advanced or metastatic solid tumors, and to preliminarily measure its anti-tumor efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary informed consent, knowledge of the study and willingness to follow and has ability to complete all trial procedures
* There is a histologically or cytologically confirmed, locally advanced or metastatic tumor by standard treatment failure or lack of standard treatment or inability to tolerate standard treatment;

For patients enrolled in the extended period:

Group 1: vascular rich tumors, including but not limited to neuroendocrine tumors, thymic squamous cell carcinoma and soft tissue Sarcoma, the specific categories are as follows. If it is necessary to enroll other types of tumor subjects, it is necessary to cooperate with the sponsor The responsible person shall discuss and confirm.

* Neuroendocrine tumor (net): low and medium grade (G1 or G2) confirmed by histopathology: low grade Other (G1) was defined as mitotic image number < 2 / 10, high power field of view [HPF] and / or Ki-67 differentiation Index < 3%; The intermediate level (G2) is defined as the number of mitotic images 2-20 / 10 high-power field of vision[HPF] and / or Ki-67 differentiation index 3-20%. If the mitotic image and Ki of the same tumor tissue-67 indicators correspond to different levels and follow higher levels;
* Thymic squamous cell carcinoma (TSCC): thymic squamous cell carcinoma confirmed by histology or cytology;
* Soft tissue sarcoma (STS): soft tissue sarcoma confirmed by histology or cytology;

Group 2: hepatocellular carcinoma (HCC): hepatocellular carcinoma confirmed histologically or cytologically. Barcelona Clinic Liver cancer stage B and C (BCLC B and C)

* The eastern United States cooperative tumor group (ECOG) score was 0 or 1
* Expect to survive at least 3 months
* Must have at least one assessable lesion as defined in RECIST v1.1;
* Suitable organs and hematopoietic function should be available. Laboratory tests during screening should meet the appropriate criteria:
* Male and female subjects of childbearing age will agree to use effective, investigator-approved contraceptive methods from the date of the informed consent until 3 months after the last administration
* Previous treatment of subjects enrolled in the extended study:
* Net: Net subjects with disease progression after at least 2-wire system antitumor drug treatment regimen: connected Systematic treatment for unresectable net, followed by recurrence / progression, or intolerance, or Unwilling to receive treatment. Frontline treatment may include somatostatin analogues, interferon, PRRT (peptide) Receptor radionuclide therapy), mTOR inhibitor or chemotherapy (unlimited chemotherapy drugs and times, Chemotherapy is regarded as a drug treatment regimen), anti angiogenesis drugs (including anti VEGF-A monoclonal antibody) Or VEGFR tyrosine kinase inhibitor);
* Thymic squamous cell carcinoma and soft tissue sarcoma: failure of previous conventional systemic chemotherapy;
* HCC: HCC subjects with disease progression or intolerance after treatment with 2-line system antitumor drugs: after receiving systematic treatment for unresectable HCC, they relapse / progress, or are unable to tolerate Those who are affected or unwilling to receive treatment. Frontline systemic therapy must include immune checkpoint inhibitors and anti-inflammatory drugs Angiogenesis drugs (including anti-vegf-a monoclonal antibody or VEGFR tyrosine kinase inhibitor).

Exclusion Criteria:

* Had suffered from malignant tumors other than the primary tumor at the time of enrollment within 5 years before screening (except: after Fully treated cervical carcinoma in situ, local squamous cell carcinoma of the skin, basal cell carcinoma, localized cancer Adenocarcinoma, ductal carcinoma in situ or stage I uterine cancer);
* High grade (G3) neuroendocrine carcinoma, adenoid carcinoma, islet cell carcinoma, goblet cell carcinoid, large Cellular neuroendocrine carcinoma and small cell carcinoma;
* Functional net and need to be accompanied by the use of long-acting somatostatin analogues to control symptoms, such as insulinoma Gastrinoma, glucagon tumor, somatostatin tumor, adrenocorticotropic hormone tumor, vascular activity Intestinal peptidoma with carcinoid syndrome, zoai syndrome or disease-specific active symptoms-
* Patients with symptoms of brain or pia meningeal metastases.
* The lung metastasis of the tumor has a cavity, or the investigator judges that there is bleeding tendency or bleeding risk;
* patients requiring local treatment or repeated drainage, the investigator identified poorly controlled effusion of the body cavity (pleural fluid, ascites, pericardial effusion, etc.)
* The adverse reactions of previous treatment did not recover to CTCAEv5.0 score ≤1 (excluding hair loss and anemia);
* Had received any previous systemic therapy targeting VEGF or VEGFR2 signaling pathway;
* Drugs or chemotherapy or radiotherapy received in other clinical trials within 4 weeks prior to enrollment (mitomycin C and nitrosorea should be administered at least 6 weeks before the last dose)
* Patients who had major surgery within 4 weeks prior to screening (excluding needle biopsy) and who were expected to have major surgery during the study period (including the 28-day screening period) or had severe unhealed wounds, ulcers, or trauma
* Left ventricular ejection fraction ≤50%;
* Heart failure patients with greater than or equal to Ⅱ level（NYHA）;
* Clinically significant arrhythmias (including frequent ventricular premature beats, symptomatic or treatable ventricular tachycardia, and asymptomatic persistent ventricular tachycardia);
* After regular antihypertensive treatment for 4 weeks, the blood pressure did not reach systolic blood pressure < 150mmhg and / or diastolic blood pressure < 150mmhg 90mmHg, or after regular antihypertensive treatment, the blood pressure reaches systolic blood pressure < 150mmhg and / or diastolic blood pressure The duration of pressure < 90mmHg is less than 4 weeks
* There are currently venous thromboemboli that require treatment;
* Myocardial infarction, stroke or other severe arterial thromboembolism events occurred within 6 months before enrollment.
* Any grade 2 or more bleeding occurred within 6 months prior to enrollment;
* Intraperitoneal abscess, or abdominal wall fistula, gastrointestinal perforation, or a history of poorly controlled/recurrent inflammatory bowel disease (including crohn's disease or ulcerative colitis) occurred within 6 months prior to enrollment.
* The patient is receiving （NSAIDS;Such as indomethacin, ibuprofen, naproxen or similar drugs) or antiplatelet drugs (such as clopidogrel, ticlopidine, dipyridamole or analgrel) for long-term treatment;Aspirin is permitted with a maximum dose of 325 mg per day;Celecoxib is permitted for analgesic treatment;However, low-dose aspirin (≤325mg/d) and celecoxib should not be used at the same time.
* Patients are known to be allergic to MSB0254 or its excients, monoclonal antibodies, or any other therapeutic protein, such as fresh frozen plasma, human serum albumin (HSA), cytokines, or interleukin.If severe allergic reactions are suspected (CTCAE v5.0 grade ≥3), the patient should be excluded.
* Urine protein concentration of patients according to dipstick or routine urine analysis (UA) is >1 +,The patients also had edema or serum albumin levels below the lower limit of the normal range (LLN).Alternatively, if the urine protein concentration of the patient is ≥2+ according to the dipstick or routine urine analysis, the urine protein concentration in the 24-hour urine protein analysis must be>1g, accompanied by edema or serum albumin lower than LLN;
* Patients with a known history of hepatitis c or chronic active hepatitis b. Except for HBV carriers, hepatitis b patients who are stable after drug treatment (hbv-dna titer must not be higher than 1000 copies [CPS]/mL or 200 IU/mL) and hepatitis c patients who are stable after drug treatment (hcv-rna negative)
* A known history of HIV infection or a positive test for human immunodeficiency virus (HIV);
* Positive treponema pallidum test;
* A history of alcohol, drug or substance abuse in the past 1 year;
* Has a clear history of neurological or mental disorders, such as epilepsy or dementia;
* Poor compliance of the subject;
* Women who are pregnant (confirmed by a urine or serum pregnancy test) or breast-feeding;
* the investigators concluded that the study was not suitable for participants for other reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of MSB0254 | Up to 90 days following the last dose
  Measured by number adverse events that are related to treatment
Maximum tolerated dose(MTD) or recommended phase2 dose（RP2D） | Up to 90 days following the last dose
  Measured by number of subjects experiencing DLT in each escalation cohort

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) for MSB0254 | Up to 30 days following the last dose
  Changes in AUC over time in subjects with MSB0254
Peak Plasma concentration (Cmax)for MSB0254 | Up to 30 days following the last dose
  Cmax is the maximum observed plasma concentration
Time to the Maximum Observed Plasma Concentration (Tmax) | Up to 30 days following the last dose
  Tmax is the time in hours/days to reach Cmax following dosing
Terminal elimination half-life (t1/2) | Up to 30 days following the last dose
  The time required for the plasma level of the study drug to decrease by one-half during the terminal elimination phase
The immunogenicity of MSB0254 injection | Up to 30 days following the last dose
  The immunogenicity of MSB0254 injection was evaluated by testing the production of anti-drug antibody (ADA).
Objective response rate (ORR) as measured by RESISTv1.1 | Up to 90 days following the last dose
  Objective response rate (ORR) as measured by RESISTv1.1
Duration of response (DOR) as measured by RESISTv1.1 | Up to 90 days following the last dose
  Duration of response (DOR) as measured by RESISTv1.1
Progression-free survival (PFS) as measured by RESISTv1.1 | Up to 90 days following the last dose
  Progression-free survival (PFS) as measured by RESISTv1.1

CONTACTS AND LOCATIONS:
Overall Officials: Mengde Wang, Study Director — Suzhou Transcenta Therapeutics Co., Ltd.
Locations (2):
- China (2):
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - FuDan University ZhongShan Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No